CLINICAL TRIAL: NCT05641714
Title: The Reliability and Validity of the L-test in Patients With Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Kader Eldemir, Research Assistant, Ordu University
Other Study IDs: 1-MS-L-Test-reliability
Record Dates: First submitted 2022-11-24; First posted 2022-12-08 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Multiple Sclerosis
Keywords: L test; multiple sclerosis; functional mobility; reliability; validity
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- multiple sclerosis: Patients with Multiple Sclerosis
  Interventions: Other: L test; Other: Timed Up and Go test; Other: 10 meter walk test; Other: Six Minute Walk Test; Other: The timed 360° turn test
- healthy controls: healthy controls
  Interventions: Other: L test

INTERVENTIONS:
Other: L test — The test includes standing up from a chair, walking in a straight line for 3 m, turning to the right, walking in a straight line for 7 m, turning around, walking back 7 m along the same line, turning to the left, walk 3 m in a straight line to the chair, and then sit down.
Other: Timed Up and Go test — The test requires the individual to stand up from an armed chair, walk 3m, turn around, walk back to the armed chair, and sit down again.
  Groups: multiple sclerosis
Other: 10 meter walk test — In the test, the clinician measures the time taken to walk a distance of 10 m from a standing position. Participants are asked to walk along a 14 m long walkway.
  Groups: multiple sclerosis
Other: Six Minute Walk Test — This test measures the distance (in m) that an individual is able to walk at a comfortable speed for 6 minutes. Starting from a standing position, participants walk continuously around two pylons placed 30 m apart for 6 minutes. The distance is recorded end of the test.
  Groups: multiple sclerosis
Other: The timed 360° turn test — Each participant turns around in place in a standing position for both sides.
  Groups: multiple sclerosis

SUMMARY:
Walking safely inside or outside is an important function in patients with Multiple Sclerosis (PwMS) that affects their daily life activity and participation. Loss of functional mobility is the major component of walking disorders in PwMS. Therefore, it is important to evaluate functional mobility.

Many functional mobility tests have been used for PwMS; however, these tests generally focus on walking speed and endurance. On the other hand, the L test, a variation of the timed up and go test (TUG), is a functional mobility measurement tool that extends the total walking distance to 20 meters and also requires the patients to turn both clockwise and counterclockwise.

Although L the test is an easy-to-use, short-term test method that evaluates higher-level components of functional mobility such as turns and transfers, to our knowledge, no study has systematically examined the reliability and validity of the L test in PwMS yet. In addition, the cut-off times that best discriminate PwMS from healthy people and fallers with non-fallers with Multiple Sclerosis (MS) have not been reported. Therefore, this study planned to investigate the reliability, validity, and discrimination of the L test in PwMS.

DETAILED DESCRIPTION:
At baseline, the L test, Timed Up and Go test, 10 meter walk test, six minute walk test, and the timed 360 turn test will be applied to the Multiple Sclerosis group. The L test will be repeated after seven days after the first application in PwMS. Healthy controls are going to perform only the L test.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 18 years,
* Neurologist-diagnosed Multiple Sclerosis,
* Expanded Disability Status Scale (EDSS) score between 0-5,
* No MS exacerbation within the last 3 months,
* Use of stable medication in the last 3 months.

Exclusion Criteria:

* Having any vision, hearing, or perception problems that may affect the research results,
* Having an orthopedic problem that will prevent walking and standing
* Having a cardiovascular, pulmonary, or hormonal disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Multiple Sclerosis who apply to Gazi University, Department of Physiotherapy and Rehabilitation will be invited to this study.
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2022-12-15 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
L test | baseline
  The L test evaluates functional mobility. Higher durations indicate worse functional mobility performance.
L test-second assessment | the second assessment will be conducted after the seven days
  The L test evaluates functional mobility. Higher durations indicate worse functional mobility performance.

SECONDARY OUTCOMES:
Timed Up and Go test | Baseline
  Timed Up and Go test evaluates functional mobility. Higher durations indicate worse functional mobility.
10 meter walk test | Baseline
  10 meter walk test is a performance measure used to assess walking speed in meters per second over a short distance. It can be employed to determine functional mobility and gait.
6 minute walk test | Baseline
  This test measures the distance (in m) that an individual is able to walk at a comfortable speed for 6 minutes. Starting from a standing position, participants walk continuously around two pylons placed 30 m apart for 6 minutes. The distance is measured end of the test.
the timed 360° turn test | Baseline
  The timed 360° turn test is an easily administered, not time-consuming, and specific measurement tool to assess turning ability. It measures the time taken for an individual to 360° turn around in a standing position. The timed 360° turn test is also correlated with balance and functional mobility.

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim JS, Chu DY, Jeon HS. Reliability and validity of the L test in participants with chronic stroke. Physiotherapy. 2015 Jun;101(2):161-5. doi: 10.1016/j.physio.2014.09.003. Epub 2014 Oct 28. PMID 25555897
- [Background] Deathe AB, Miller WC. The L test of functional mobility: measurement properties of a modified version of the timed "up & go" test designed for people with lower-limb amputations. Phys Ther. 2005 Jul;85(7):626-35. PMID 15982169
- [Derived] Eldemir K, Eldemir S, Ozkul C, Irkec C, Guclu-Gunduz A. Reliability and validity of the L test in people with multiple sclerosis. Physiotherapy. 2025 Mar;126:101429. doi: 10.1016/j.physio.2024.101429. Epub 2024 Sep 24. PMID 39541755